CLINICAL TRIAL: NCT00138333
Title: Assessment of Mercury Levels and Metabolism in Premature and Low Birth Weight (LBW) Infants Receiving Vaccines Containing Thimerosal
Brief Title: Mercury Levels in Premature and LBW Infants Receiving Thimerosal-containing Vaccines
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Other Study IDs: 04-046
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2007-10

CONDITIONS: Mercury Levels
Keywords: Thimerosal, mercury levels, low birth weight, Argentina

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The goal of the study is to find out how much mercury is in the blood, urine, and stools of premature and low birth weight infants who have received standard childhood vaccines that are given to all infants in Argentina. Seventy-two newborn premature and low birth weight infants from Durand Acute General hospital will participate in this study. Each infant in the study will need to make two visits, one at the time of vaccination and another 12 hours to 30 days later. Urine, stool, and a small sample of blood will be taken at each visit.

DETAILED DESCRIPTION:
The primary objective is to describe the levels of mercury in the blood of premature newborns greater than or equal to 32 weeks and less than 37 weeks gestation and birth weight greater than or equal to 2000 grams but less than 3000 grams, who receive the routine birth dose of Hepatitis B immunization containing ethyl mercury in the form of thimerosal and the birth dose of BCG immunization, and to evaluate the excretion of mercury in these newborns by examining mercury levels in stool and urine. Secondary objectives are: 1) to determine the half-time of mercury in blood following vaccination of premature and low birth weight infants with thimerosal-containing vaccines, and 2) to screen premature and low birth weight infants for evidence of early effects of thimerosal on the kidney by measurement of urinary gamma glutamyl transpeptidase levels. All infants will have stool, urine, and blood samples collected prior to receipt of routine birth hepatitis B and BCG immunization. Cord blood will serve as the baseline blood specimen. Each infant will be seen once at a predetermined follow-up visit time point. There will be 6 follow-up visit time points, with sampling from 12 infants at each time point. All infants will provide blood, urine, and stool specimens at the assigned follow-up visit.

ELIGIBILITY:
Inclusion Criteria: 1) Parent/guardian gives written informed consent. 2) Good health as determined by negative gestational history, subject's medical history and physical assessment. Medical history will include a review of the major body systems (e.g., ear-nose-throat, cardiovascular, respiratory, neurological, gastrointestinal, genitourinary, hematological). 3) Newborn cohort: within 3 days of birth and gestational age = 32 weeks and < 37 weeks and a birth weight = 2000 grams and < 3000 grams. 4) Able to attend the scheduled visits and to comply with the study procedures. Exclusion Criteria: 1) Infant history of vaccinations and date received is unknown or undocumented. 2) Known history of high-level mercury exposure in mother or infant. 3) Any contraindication to routine vaccinations. 4) Clinically significant findings on review of systems (determined by investigator or sub-investigator to be sufficient for exclusion). 5) Known or suspected impairment of immunologic function or receipt of immunosuppressive therapy or immunoglobulin since birth. 6) HIV-positive mother by history. 7) Personal or immediate family history of congenital immune deficiency. 8) Developmental delay or neurological disorders.

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2005-12; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Ninos, "Ricardo Gutierrez", Buenos Aires, Argentina